CLINICAL TRIAL: NCT05843890
Title: Tailored Pain Guide (TPG) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Daniel Clauw, MD, Professor of Anesthesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00214375
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lower Back Pain
Keywords: Online resources; Fitbit; Surveys

STUDY DESIGN:
Intervention Model Description: The initial study enrolled 297 participants. Following the amendment (AME00158411) the study team will now enroll the non-pharma program to this project. The anticipated enrollment number was increased from 430 to 550.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Structured and tailored PainGuide (Experimental)
  Interventions: Behavioral: Structured and tailored PainGuide
- Standard PainGuide (Active Comparator)
  Interventions: Behavioral: Standard PainGuide

INTERVENTIONS:
Behavioral: Structured and tailored PainGuide — Participants will receive specific instruction to complete one module a week over the first 4 weeks. Participants will then receive tailored messaging using scores from the assessments completed during T1(baseline visit) from the PROMIS 29+2.
  The initial group of participants (prior to AME00158411) will complete surveys for 24 weeks.
  The NPP Participants will be asked to complete surveys for 52 weeks.
  All participants will also be registered with a Fitbit device that is linked to the PainGuide to capture movement data (daily step counts).
  Arms: Structured and tailored PainGuide
Behavioral: Standard PainGuide — Participants in the control group will not receive any messaging once enrolled. The initial group of participants (prior to AME00158411) will complete surveys for 24 weeks.
  The NPP Participants will be asked to complete surveys for 52 weeks.
  All participants will also be registered with a Fitbit device that is linked to the PainGuide to capture movement data (daily step counts).
  Arms: Standard PainGuide

SUMMARY:
This research is studying whether changing an individual's behaviors may have an impact as a treatment or outcome for chronic low back pain. This research will try to understand how much an electronic, self-management website like PainGuide can help participants.

The study hypothesizes that tailored digital interventions (plus using PainGuide) will demonstrate greater improvement in pain interference.

DETAILED DESCRIPTION:
There was an amendment approved by the University of Michigan Medical School Institutional Review Board (AME00158411). This amendment included the following:

increased enrollment numbers, updated recruitment procedures including the Non-Pharma Program (NPP) Sub-Study, as well as changes in time frames.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Lower Back pain (cLBP) defined by the National Institutes of Health (NIH) Task Force Report on Research Standards for Chronic Low Back Pain, (i.e., low back pain present at least six months, and present more than half of those days.)
* Individuals must have a score of greater or equal to (≥) 60 on PROMIS Pain Interference.
* Non-Pharma Sub-study:

  1. Must be referred and currently on the waitlist for the NPP at the Back & Pain Center (BPC)

Exclusion Criteria:

* Current cancer related pain
* Diagnosis of autoimmune disease
* Unable to speak, write or read English
* Visual or hearing difficulties
* Pregnancy or breastfeeding
* Any other diseases or conditions that would make a patient unsuitable for study participation as determined by the site principal investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference score | Baseline, Week 24
  The PROMIS Pain Interference consists of 4-items that assess the degree to which pain interferes with various aspects of life. Items are scored on a 1 ("Not at all") to 5 ("Very much") scale with a range of 4 - 20. Higher scores indicate greater pain interference

SECONDARY OUTCOMES:
Change in pain intensity based on the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 version 2.0 | Baseline, Week 24 (initial group), Week 52 (NPP group)
  There is one question that participants select 0 (no pain) - 10 (worst imaginable pain).
Change in the Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive function | Baseline, Week 24 (initial group), Week 52 (NPP group)
  There are 2 questions regarding cognitive function where participants select answers from not at all (1)-very mush (5) regarding cognitive function. There is a total of 10 points where higher scores mean higher cognitive function.
Change in the physical function based on the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 version 2.0 | Baseline, Week 24 (initial group), Week 52 (NPP group)
  There are 4 questions that participants will select from without any difficulty (5) to unable to do (1). There are a total of 20 points where higher scores indicate higher physical function.
Change in anxiety based on the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 version 2.0 | Baseline, Week 24 (initial group), Week 52 (NPP group)
  There are 4 questions that participants will select from never (1) to always (5). There are a total of 20 points where lower scores indicate lower levels of anxiety.
Change in depression based on the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 version 2.0 | Baseline, Week 24 (initial group), Week 52 (NPP group)
  There are 4 questions that participants will select from never (1) to always (5). There are a total of 20 points where higher scores indicate higher levels of depression.
Change in fatigue based on the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 version 2.0 | Baseline, Week 24 (initial group), Week 52 (NPP group)
  There are 4 questions that participants will select from not at all (1) to very much (5). There are a total of 20 points where higher scores indicate higher levels of fatigue.
Change in sleep disturbance based on the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 version 2.0 | Baseline, Week 24 (initial group), Week 52 (NPP group)
  There are 4 questions that participants will select from. Question 1 participants will select from Very poor (5) to very good. Questions 2-4 participants will select from not all (5) to very much (1). There are a total of 20 points where higher scores indicate higher sleep disturbances.
Change in ability to participate in social roles and activities based on the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 version 2.0 | Baseline, Week 24 (initial group), Week 52 (NPP group)
  There are 4 questions that participants will select from never (5) to always (1). There are a total of 20 points where lower scores indicate more difficulty participating in social roles.
Change in pain interference based on the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 version 2.0 | Baseline, Week 24 (initial group), Week 52 (NPP group)
  There are 4 questions that participants will select from not at all (1) to very much (5). There are a total of 20 points where lower scores indicate less pain interference.
Change in pain interference based on the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 version 2.0 - between baseline and 52 weeks for NPP participants | Baseline, Week 52 (T5)
  There are 4 questions that participants will select from not at all (1) to very much (5). There are a total of 20 points where lower scores indicate less pain interference.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Clauw, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No